CLINICAL TRIAL: NCT04852770
Title: A Randomized Clinical Trial to Assess the Efficacy of Online Treatment With Trial-based Cognitive Therapy, Mindfulness-based Health Promotion and Positive Psychotherapy for Post-traumatic Stress Disorder During the Covid-19 Pandemics
Brief Title: Efficacy of TBCT, MBHP and PPT for PTSD During the Covid-19 Pandemics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was interrupted due to the end of the pandemic.
Sponsor: Fundação Bahiana de Infectologia (Other)
Collaborators: Mente Aberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FundacaoBI
Record Dates: First submitted 2020-12-22; First posted 2021-04-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder; Covid19
Keywords: Cognitive-Behavior Therapy; Trial-Based Cognitive Therapy; Mindfulness Based Health Promotion; Positive Psychotherapy; PTSD; Covid 19; Randomized clinical trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Trial-Based Cognitive Therapy (Experimental): TBCT (de Oliveira, 2008) is a novel transdiagnostic approach (Wenzel, 2017). It has been shown to be effective for depression (Hemanny et al., 2019), social anxiety disorder (Neufeld et al., 2020; Caetano et al., 2018; de Oliveira et al., 2011; Powell et al., 2013), and PTSD (Duran et al., 2020). TBCT differs from other CBT approaches in that it introduces a new, organized, and systematic approach to change dysfunctional negative core beliefs, and allows cognitive, emotional, and experiential work to be done simultaneously (de Oliveira, 2016). Interestingly, it incorporates a courtroom metaphor to challenge dysfunctional core beliefs conceptualized as self-accusations (de Oliveira, 2016). TBCT is an example of assimilative psychotherapy integration that relies on Beckian CBT (de Oliveira, 2016). It incorporates and integrates components of other psychotherapies (Delavechia et al., 2016).
  Interventions: Behavioral: Trial-Based Cognitive Therapy
- Mindfulness-Based Health Promotion (Active Comparator): The Mindfulness-Based Stress Reduction (MBSR) program was created by Jon Kabat-Zinn and colleagues at the University of Massachusetts Medical Center in 1979, and it is an intervention whose effects on mental health and quality of life has produced several studies worldwide, both in clinical and non-clinical populations. Several protocols have been developed based on the MBSR aimed at specific publics, such as the Mindfulness-Based Health Promotion (MBHP) program developed by the Mente Aberta - Brazilian Center for Mindfulness and Health Promotion. The MBHP program was inspired by the original MBSR model but adapted to the context of the Brazilian Health Care (SUS) system, addressing chronic conditions and mental disorders as well (TROMBKA et al., 2018; LOPES et al., 2019; SALVO et al., 2018).
  Interventions: Behavioral: Mindfulness-Based Health Promotion
- Positive psychotherapy (Active Comparator): Positive psychotherapy (PPT) seeks to understand positive emotions, psychological potentialities and healthy human / social / institutional functioning, and to apply this knowledge to help people and institutions, with a focus on prevention and promotion of mental health (SELIGMAN et al., 2005). Originally, PP focused on happiness and subjective well-being (SELIGMAN, 2010; SELIGMAN; CSIKSZENTMIHALYI, 2000). Then, the studies gained a broader view of psychological well-being and another similar proposal entitled PERMA, which is composed of the following five spheres: positive emotions - P; engagement - E; relationships - R; meaning - M; and achievement - A. (RYFF, 2013; SELIGMAN, 2012). Although positive psychology aims to be a way of looking at life, some psychotherapeutic proposals, such as positive psychotherapy (PPT), have been developed, and clinical studies have been replicated in different clinical and cultural contexts (RASHID; SELIGMAN, 2019; RICHES et al., 2016).
  Interventions: Behavioral: Positive psychotherapy

INTERVENTIONS:
Behavioral: Trial-Based Cognitive Therapy — TBCT is an approach that includes psychoeducation and cognitive restructuring techniques concerning automatic thoughts, underlying assumptions and core beliefs related to the traumatic events. It is conducted in a therapeutic setting that makes use of experiential techniques, allowing the patient to refer to him/herself in the third person and thus taking distance from him or herself. One of TBCT techniques for dealing with guilt and shame, emotions that provoke great limitation to patients with PTSD, is the participation grid (PG). Another important technique is the consensual role-play (CRP), designed to help patients resolve ambivalence and make decisions. In addition, the most important TBCT technique, the Trial, was developed to help patients change dysfunctional negative core beliefs. Therapists who will conduct this approach have a specialization level in CBT. In this study, this treatment will be delivered in 14 sessions, weekly, individualy, one session by week and on line.
  Other Names: TBCT
  Arms: Trial-Based Cognitive Therapy
Behavioral: Mindfulness-Based Health Promotion — The MBHP protocol is a structured program developed over 8 sessions, in group, where participants (8-15 people) meet every week for 2 hours (standard duration of one session), to experience the concepts and techniques of mindfulness. Participants are also given suggestions of daily activities to be implemented at home or in the workplace, that last in average 15-20 minutes, but may last up to 45 minutes in the case of more motivated and compliant participants. They are also encouraged to incorporate the idea of Mindfulness in their daily lives (the so-called "informal practice"), so that all daily activities somehow become opportunities to practice Mindfulness. In this study, this treatment will be delivered in 14 sessions, weekly, individualy, one session by week and on line.
  Other Names: MBHP
  Arms: Mindfulness-Based Health Promotion
Behavioral: Positive psychotherapy — PPT is the clinical and therapeutic work derived from PP. PPT consists of 15 specific practices that have been empirically validated, either separately, or in conjunction with two or three practices. After empirical validation, these practices were organized in a cohesive protocol of 15 sessions called PPT. Many of these practices have been studied through online interventions. In the present study, the protocol will be reduced to 14 sessions, with sessions called positive relationships, positive communication, and practical wisdom removed. It was understood that the other 12 would be more easily adapted to the moment of the study. (DUCKWORTH; STEEN; SELIGMAN, 2005; MONGRAIN; ANSELMO-MATTHEWS, 2012; RASHID; SELIGMAN, 2019). In this study, this treatment will be delivered in 14 sessions, weekly, individualy, one session by week and on line.
  Other Names: PPT
  Arms: Positive psychotherapy

SUMMARY:
The psychotherapies to be assessed in the present study, delivered on-line, are: trial-based cognitive therapy (TBCT), mindfulness-based health promotion (MBHP), and positive psychotherapy (PPT). Objectives: 1) to assess the efficacy of TBCT compared to MBHP and PPT in reducing the symptoms of PTSD during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Background: Research has suggested the use of different forms of psychotherapy to decrease drop-out rates in the post-traumatic stress disorder (PTSD) treatment. The psychotherapies to be assessed in the present study are: trial-based cognitive therapy (TBCT), mindfulness-based health promotion (MBHP) and Positive psychotherapy (PPT). Objectives: Our objectives are: 1) to assess the efficacy of TBCT compared to MBHP and PPT to reduce the symptoms of PTSD in the context of the COVID-19 pandemic, all delivered online; 2) to compare the efficacy of these psychotherapies in reducing symptoms of anxiety and depression, and in improving well-being; 3) to describe how patients and professionals perceive teletherapy. Methods: This is a three-arm, randomized, multicenter, single-blind, clinical trial. An estimated sample of 135 patients will receive either TBCT, MBHP or PPT, individual, weekly visits, totaling thirteen sessions. The primary outcome measure will be the CAPS-5, and the secondary outcome measures will be the Hospital Anxiety and Depression Scale (HADS), the Negative Core Beliefs Inventory (NCBI), and the Trauma-Related Guilt Inventory (TRGI). Other measures are the WHO-5 Well-being Index (WHO-5), and the California Psychotherapy Alliance Scale (CALPAS-P). Also, questions about patients perception of teletherapy will be asked. Expected results: PTSD symptoms are expected to be reduced after TBCT, MBHP and PPT. The null hypothesis is that no statistical difference is expected to be found among the three psychotherapies, as opposed to the alternative hypothesis that TBCT and MBHP are superior to PPT.

ELIGIBILITY:
Inclusion criteria:

* both sexes;
* aged 18 to 60 years;
* scoring 45 or more on the PCL-5
* PTSD developed (or aggravated by) as a result of direct or indirect exposure to COVID-19 [e.g., health professionals, people who tested positive for Covid-19 (or their relative or close friends), or those who quarantined, isolated or socially distanced themselves];
* Participants should be able to read, write and follow instructions, and have access to the a stable internet connexion.

Exclusion Criteria:

* severe suicide risk (plans, attitudes or suicide attemps for the last 12 months);
* self-mutilation behavior (for the last 12 months);
* already in psychotherapy;
* psychotic symptoms;
* current substance abuse or addiction (last 12 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
The Clinician-Administered PTSD Scale (CAPS-5) | Baseline and week 14.
  It is a diagnostic interview scale with 30 items to assess the diagnosis and the severity of PTSD symptoms according to DSM-5 (Weathers et al., 2018)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline and week 14.
  This is a fourteen-item scale used to assess anxiety and depression symptoms, where each item scores 0 to 3 points, and a total score of 9 or higher suggests mild symptoms. It was translated and validated for the Brazilian population. (Faro, 2015; Zigmond e Snaith, 1983).
Hospital Anxiety and Depression Scale (HADS) | From baseline to post-treatment, up 14 weeks.
  This is a fourteen-item scale used to assess anxiety and depression symptoms, where each item scores 0 to 3 points, and a total score of 9 or higher suggests mild symptoms. It was translated and validated for the Brazilian population. (Faro, 2015; Zigmond e Snaith, 1983).
Trauma-Related Guilt Inventory (TRGI) | Baseline and week 14.
  This is a 32-item questionnaire assessing the cognitive and emotional aspects of guilt which are associated to a specific traumatic event.
Negative Core Beliefs Inventory (NCBI) | Baseline and week 14.
  Designed to assess negative core beliefs, as described by Beck (2005); it consists of 50 items evaluating beliefs about oneself and other people, on a likert scale of 1 to 4 points each (Osmo, 2017).
The World Health Organization Five Well-being index (WHO-5) | Baseline and week 14.
  Overall well-being scale, with five questions and scores ranging from 0-5, addressing mood and energy (TOPP et al., 2015; DADFAR, 2018). The WHO-5 validation study into Brazilian Portuguese included 1,128 individuals. In this study, the instrument presented good internal validity (Cronbach's alpha = 0,83)
California Psychotherapy Alliance Scale - Patient version (CALPAS-P) | From baseline to post-treatment, up to 14 weeks.
  It is a scale that assess four components of therapeuthic alliance: work, relation, comprehension of therapist and objectives of treatment for the patient.

OTHER OUTCOMES:
Structured Clinical Interview for DSM-5 - SCID | Baseline
  It is a semi-structured psychiatric interview, with the purpose of providing a diagnosis, according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
Posttraumatic stress disorder checklist for DSM-5 (PCL-5) | Baseline.
  It contains 20 items with the purpose of assessing PTSD symptoms, in accordance with criteria B, C, D and E (DSM-5). Each item is scored in a scale that ranges from 0 (not at all) to 4 (extremely).
The Clinician-Administered PTSD Scale (CAPS-5) | Week 7.
  It is a diagnostic interview scale with 30 items to assess the diagnosis and the severity of PTSD symptoms according to DSM-5 (Weathers et al., 2018)
The Clinician-Administered PTSD Scale (CAPS-5) | 6 months.
  It is a diagnostic interview scale with 30 items to assess the diagnosis and the severity of PTSD symptoms according to DSM-5 (Weathers et al., 2018)
The Clinician-Administered PTSD Scale (CAPS-5) | 12 months.
  It is a diagnostic interview scale with 30 items to assess the diagnosis and the severity of PTSD symptoms according to DSM-5 (Weathers et al., 2018)
The Clinician-Administered PTSD Scale (CAPS-5) | 18 months.
  It is a diagnostic interview scale with 30 items to assess the diagnosis and the severity of PTSD symptoms according to DSM-5 (Weathers et al., 2018)
Hospital Anxiety and Depression Scale (HADS) | Week 7.
  This is a fourteen-item scale used to assess anxiety and depression symptoms, where each item scores 0 to 3 points, and a total score of 9 or higher suggests mild symptoms. It was translated and validated for the Brazilian population. (Faro, 2015; Zigmond e Snaith, 1983).
Hospital Anxiety and Depression Scale (HADS) | 6 months
  This is a fourteen-item scale used to assess anxiety and depression symptoms, where each item scores 0 to 3 points, and a total score of 9 or higher suggests mild symptoms. It was translated and validated for the Brazilian population. (Faro, 2015; Zigmond e Snaith, 1983).
Hospital Anxiety and Depression Scale (HADS) | 12 months
  This is a fourteen-item scale used to assess anxiety and depression symptoms, where each item scores 0 to 3 points, and a total score of 9 or higher suggests mild symptoms. It was translated and validated for the Brazilian population. (Faro, 2015; Zigmond e Snaith, 1983).
Hospital Anxiety and Depression Scale (HADS) | 18 months
  This is a fourteen-item scale used to assess anxiety and depression symptoms, where each item scores 0 to 3 points, and a total score of 9 or higher suggests mild symptoms. It was translated and validated for the Brazilian population. (Faro, 2015; Zigmond e Snaith, 1983).
Trauma-Related Guilt Inventory (TRGI) | Week 7.
  This is a 32-item questionnaire assessing the cognitive and emotional aspects of guilt which are associated to a specific traumatic event.
Trauma-Related Guilt Inventory (TRGI) | 6 months.
  This is a 32-item questionnaire assessing the cognitive and emotional aspects of guilt which are associated to a specific traumatic event.
Trauma-Related Guilt Inventory (TRGI) | 12 months.
  This is a 32-item questionnaire assessing the cognitive and emotional aspects of guilt which are associated to a specific traumatic event.
Trauma-Related Guilt Inventory (TRGI) | 18 months.
  This is a 32-item questionnaire assessing the cognitive and emotional aspects of guilt which are associated to a specific traumatic event.
Negative Core Beliefs Inventory (NCBI) | Week 7.
  Designed to assess negative core beliefs, as described by Beck (2005); it consists of 50 items evaluating beliefs about oneself and other people, on a likert scale of 1 to 4 points each (Osmo, 2017).
Negative Core Beliefs Inventory (NCBI) | 6 months.
  Designed to assess negative core beliefs, as described by Beck (2005); it consists of 50 items evaluating beliefs about oneself and other people, on a likert scale of 1 to 4 points each (Osmo, 2017).
Negative Core Beliefs Inventory (NCBI) | 12 months.
  Designed to assess negative core beliefs, as described by Beck (2005); it consists of 50 items evaluating beliefs about oneself and other people, on a likert scale of 1 to 4 points each (Osmo, 2017).
Negative Core Beliefs Inventory (NCBI) | 18 months.
  Designed to assess negative core beliefs, as described by Beck (2005); it consists of 50 items evaluating beliefs about oneself and other people, on a likert scale of 1 to 4 points each (Osmo, 2017).
The World Health Organization Five Well-being index (WHO-5) | Week 7.
  Overall well-being scale, with five questions and scores ranging from 0-5, addressing mood and energy (TOPP et al., 2015; DADFAR, 2018). The WHO-5 validation study into Brazilian Portuguese included 1,128 individuals. In this study, the instrument presented good internal validity (Cronbach's alpha = 0,83)
The World Health Organization Five Well-being index (WHO-5) | 6 months
  Overall well-being scale, with five questions and scores ranging from 0-5, addressing mood and energy (TOPP et al., 2015; DADFAR, 2018). The WHO-5 validation study into Brazilian Portuguese included 1,128 individuals. In this study, the instrument presented good internal validity (Cronbach's alpha = 0,83)
The World Health Organization Five Well-being index (WHO-5) | 12 months
  Overall well-being scale, with five questions and scores ranging from 0-5, addressing mood and energy (TOPP et al., 2015; DADFAR, 2018). The WHO-5 validation study into Brazilian Portuguese included 1,128 individuals. In this study, the instrument presented good internal validity (Cronbach's alpha = 0,83)
The World Health Organization Five Well-being index (WHO-5) | 18 months
  Overall well-being scale, with five questions and scores ranging from 0-5, addressing mood and energy (TOPP et al., 2015; DADFAR, 2018). The WHO-5 validation study into Brazilian Portuguese included 1,128 individuals. In this study, the instrument presented good internal validity (Cronbach's alpha = 0,83)
Semi-structured interview regarding online psychotherapy and pandemics. | Week 14.
  It consists of semi-structured questions about the perception of the patient and of the psychotherapist about the conduction of psychotherapy in an on line format, such as: quality of the therapeutic relationship and experience in on line treatment and the effect of pandemics on mental heatlh.

CONTACTS AND LOCATIONS:
Overall Officials: Irismar Reis de Oliveira, MD, PhD, Study Director — Federal University of Bahia
Locations (3):
- Brazil (3):
  - Universidade Federal da Bahia, Salvador, Estado de Bahia
  - Universidade Federal de Pernambuco, Recife, Pernambuco
  - Universidade Federal de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neufeld CB, Palma PC, Caetano KAS, Brust-Renck PG, Curtiss J, Hofmann SG. A randomized clinical trial of group and individual Cognitive-Behavioral Therapy approaches for Social Anxiety Disorder. Int J Clin Health Psychol. 2020 Jan-Apr;20(1):29-37. doi: 10.1016/j.ijchp.2019.11.004. Epub 2019 Dec 24. PMID 32021616
- [Background] Powell VB, Oliveira OH, Seixas C, Almeida C, Grangeon MC, Caldas M, Bonfim TD, Castro M, Galvao-de Almeida A, Moraes Rde O, Sudak D, de-Oliveira IR. Changing core beliefs with trial-based cognitive therapy may improve quality of life in social phobia: a randomized study. Braz J Psychiatry. 2013 Jul-Sep;35(3):243-7. doi: 10.1590/1516-4446-2012-0863. PMID 24142084
- [Background] Oliveira IR. Trial-Based Thought Record (TBTR): preliminary data on a strategy to deal with core beliefs by combining sentence reversion and the use of analogy with a judicial process. Braz J Psychiatry. 2008 Mar;30(1):12-8. doi: 10.1590/s1516-44462008000100003. PMID 18373017
- [Background] de Oliveira IR, Powell VB, Wenzel A, Caldas M, Seixas C, Almeida C, Bonfim T, Grangeon MC, Castro M, Galvao A, de Oliveira Moraes R, Sudak D. Efficacy of the trial-based thought record, a new cognitive therapy strategy designed to change core beliefs, in social phobia. J Clin Pharm Ther. 2012 Jun;37(3):328-34. doi: 10.1111/j.1365-2710.2011.01299.x. Epub 2011 Sep 28. PMID 21955037
- [Background] Hemanny C, Carvalho C, Maia N, Reis D, Botelho AC, Bonavides D, Seixas C, de Oliveira IR. Efficacy of trial-based cognitive therapy, behavioral activation and treatment as usual in the treatment of major depressive disorder: preliminary findings from a randomized clinical trial. CNS Spectr. 2020 Aug;25(4):535-544. doi: 10.1017/S1092852919001457. Epub 2019 Nov 26. PMID 31769377
- [Background] de Oliveira IR, Hemmany C, Powell VB, Bonfim TD, Duran EP, Novais N, Velasquez M, Di Sarno E, Alves GL, Cesnik JA; Brazilian TBTR Study Group. Trial-based psychotherapy and the efficacy of trial-based thought record in changing unhelpful core beliefs and reducing self-criticism. CNS Spectr. 2012 Mar;17(1):16-23. doi: 10.1017/S1092852912000399. PMID 22790114
- [Background] Duran EP, Corchs F, Vianna A, Araujo AC, Del Real N, Silva C, Ferreira AP, De Vitto Francez P, Godoi C, Silveira H, Matsumoto L, Gebara CM, de Barros Neto TP, Chilvarquer R, de Siqueira LL, Bernik M, Neto FL. A randomized clinical trial to assess the efficacy of trial-based cognitive therapy compared to prolonged exposure for post-traumatic stress disorder: preliminary findings. CNS Spectr. 2021 Aug;26(4):427-434. doi: 10.1017/S1092852920001455. Epub 2020 May 26. PMID 32450928
- [Background] Seligman MEP. Positive Psychology: A Personal History. Annu Rev Clin Psychol. 2019 May 7;15:1-23. doi: 10.1146/annurev-clinpsy-050718-095653. Epub 2018 Dec 10. PMID 30525996
- [Background] Duckworth AL, Steen TA, Seligman ME. Positive psychology in clinical practice. Annu Rev Clin Psychol. 2005;1:629-51. doi: 10.1146/annurev.clinpsy.1.102803.144154. PMID 17716102
- [Background] Mongrain M, Anselmo-Matthews T. Do positive psychology exercises work? A replication of Seligman et al. (2005). J Clin Psychol. 2012 Apr;68(4):382-9. doi: 10.1002/jclp.21839. PMID 24469930
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Trombka M, Demarzo M, Bacas DC, Antonio SB, Cicuto K, Salvo V, Claudino FCA, Ribeiro L, Christopher M, Garcia-Campayo J, Rocha NS. Study protocol of a multicenter randomized controlled trial of mindfulness training to reduce burnout and promote quality of life in police officers: the POLICE study. BMC Psychiatry. 2018 May 25;18(1):151. doi: 10.1186/s12888-018-1726-7. PMID 29801444
- [Background] de Oliveira IR. Kafka's trial dilemma: proposal of a practical solution to Joseph K.'s unknown accusation. Med Hypotheses. 2011 Jul;77(1):5-6. doi: 10.1016/j.mehy.2011.03.010. Epub 2011 Mar 31. PMID 21458165
- [Background] de Souza CM, Hidalgo MP. World Health Organization 5-item well-being index: validation of the Brazilian Portuguese version. Eur Arch Psychiatry Clin Neurosci. 2012 Apr;262(3):239-44. doi: 10.1007/s00406-011-0255-x. Epub 2011 Sep 7. PMID 21912931
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/35055641/ — Duran, É. P., Hemanny, C., Vieira, R., Nascimento, O., Machado, L., de Oliveira, I. R., & Demarzo, M. (2022). A Randomized Clinical Trial to Assess the Efficacy of Online-Treatment with Trial-Based Cognitive Therapy, Mindfulness-Based Health Promotion and Positive Psychotherapy for Post-Traumatic Stress Disorder during the COVID-19 Pandemic: A Study Protocol. International Journal of Environmental Research and Public Health, 19(2), 819.